CLINICAL TRIAL: NCT01206543
Title: Intraoperative Use of a MR Tomography System Combined With Neuronavigation - Analysis of the Craniopharyngioma Subgroup ("Intraoperative Nutzung Eines Kernspintomographie-Systems in Direkter Kopplung Mit Einem Neuronavigations-System")
Brief Title: 1.5T Intraoperative MR Imaging in Craniopharyngiomas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hofmann, Bernd, M.D. (Individual)
Responsible Party: Department of Neurosurgery, University of Erlangen-Nuremberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cranio 15
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Craniopharyngioma
Keywords: Craniopharyngioma; Surgery; Intraoperative imaging; Rate of total removal
MeSH Terms: conditions — Craniopharyngioma

ARMS (1):
- Intraoperative imaging (Experimental)
  Interventions: Other: Intraoperative imaging using 1.5T MRI

INTERVENTIONS:
Other: Intraoperative imaging using 1.5T MRI — Intraoperative imaging and determination of degree of resection / complete tumor removal

SUMMARY:
Purpose of this study is to investigate whether intraoperative imaging using a 1.5T MRI in craniopharyngioma surgery is useful in order to increase the rate of complete tumor removal.

ELIGIBILITY:
Inclusion Criteria:

* complex craniopharyngioma > 1cm extension within 2 or more cranial fossae or ventricular system
* Patient or legal representative able to provide written informed consent

Exclusion Criteria:

* tumor size< 1 cm
* Patients with any condition considered a contraindication to MRI
* Patients with any condition considered a contraindication for surgery
* Hypothalamic disturbances
* Hypothalamic edema

Ages: 3 Years to 75 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-04; Primary Completion 2005-09 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Rate of additional tumor removal | up to 3-4 months following surgery
  Number of patients in whom non suspected tumor remants were indicated by intraoperative MRI and remnants could be removed completely thereafter. Results have to be confirmed in 1st follow up imaging.
Rate of achievement of intended extent of removal | up to three months following surgery
  It is examined whether the extent of tumor removal defined prior to surgery was achieved
Diagnostic reliability | within 3 -4 months following surgery
  false positive or negative interpretation of intraoperative imaging determined after follow-up imaging 3 - 4 months following surgery

SECONDARY OUTCOMES:
Surgical complication | within 1st week following surgery
  Rate of new deficits following surgery (excluding new endocrine deficits)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Hofmann, MD, Principal Investigator
Locations (1):
- Department of Neurosurgery University of Erlangen, Erlangen, Germany